CLINICAL TRIAL: NCT03293420
Title: Retrospective Analysis of a Population of Patients With With Severe Traumatic Head Injury and Woken Early
Acronym: PRECOCE TC
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Other Study IDs: LITTEL-GIRARD 2016
Record Dates: First submitted 2017-09-21; First posted 2017-09-26 (Actual); Last update posted 2017-09-26 (Actual); Status verified 2017-09

CONDITIONS: Traumatic Head Injury

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Observational retrospective study that included all patients meeting the inclusion criteria from 1st January 2014 to 31st December 2015.

The objective of the study is to describe and compare two populations of patients with severe traumatic head injury arriving under sedation in the Department in whom the sedation was not continued.

ELIGIBILITY:
Inclusion Criteria:

- Patients with traumatic head injuring arriving in the Neurosurgery and Traumatologic Intensive Care Unit under sedation

Exclusion Criteria:

* Brain death within the 48h following admission,
* Stroke leading to the traumatic head injury,
* Death within the 24h following admission,
* Patients not under sedation on admission to the unit,
* Non-sedated patients transferred directly to the operating theatre
* Traumatic brain injury in patients presenting chronic sub-dural haematoma,
* Continued sedation (> 15h) in the ICU.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with traumatic head injury
Sampling Method: Non-Probability Sample
Enrollment: 61 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Motor score | At baseline

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Dijon Bourgogne, Dijon, France